CLINICAL TRIAL: NCT04361474
Title: A Randomized Controlled Trial Evaluating the Efficacy of Local Budesonide Therapy in the Management of Hyposmia in COVID-19 Patients Without Signs of Severity
Brief Title: Trial Evaluating the Efficacy of Local Budesonide Therapy in the Management of Hyposmia in COVID-19 Patients Without Signs of Severity
Acronym: COVIDORL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: Hopital Lariboisière (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MDL_2020_10; 2020-001667-85 (EudraCT Number)
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Budesonide; Olfaction Disorders; SARS-CoV-2; Anosmia
MeSH Terms: conditions — Olfaction Disorders; Anosmia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Patients with persistent hyposmia related to a SARS-CoV-2 infection
Who Masked: Participant
Masking Description: Patients with persistent hyposmia related to a SARS-CoV-2 infection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Nasal irrigation with budesonide and physiological saline (Budesonide 1mg/2mL diluted in 250mL of physiological saline 9°/00): 3 syringes of 20mL in each nasal cavity, morning and evening, for 30 days, in addition to olfactory rehabilitation twice a day.
  Interventions: Drug: Budesonide Nasal
- Control group (Placebo Comparator): Nasal irrigation with physiological saline 9°/00 only: 3 syringes of 20cc in each nasal cavity, morning and evening, for 30 days, in addition to olfactory re-education twice a day.
  Interventions: Other: Physiological serum

INTERVENTIONS:
Drug: Budesonide Nasal — Nasal irrigation with budesonide and physiological saline morning and evening, for 30 days, in addition to olfactory rehabilitation twice a day.
  Other Names: Experimental group
  Arms: Experimental group
Other: Physiological serum — Nasal irrigation with physiological saline morning and evening, for 30 days, in addition to olfactory re-education twice a day.
  Other Names: Control group
  Arms: Control group

SUMMARY:
The initial symptoms described in the first cases of COVID-19 were mainly fever and respiratory signs. Recently, there has been an increase in cases of hyposmia without associated nasal obstruction or rhinorrhea. Although we do not yet know the long-term consequences of COVID-19 on olfaction, there is evidence in the literature demonstrating that post-viral hyposmias are an important source of long-term olfactory disorders, impacting quality of life.

Usually, the treatment of viral hyposmias is based on local and/or general corticosteroid treatment combined with saline nasal irrigation at the onset of signs. Because of the possible development of severe forms of the SARS-Cov-2 infection, the French Society of Otorhinolaryngology has advised against treatment by corticosteroid therapy and nasal irrigation. However, as the virus is present in the nasal fossae on average for 20 days, persistent hyposmia at 30 days would probably result from an inflammatory or neurological damage to the nasal slits or olfactory bulb. Local treatment with corticosteroids could then be instituted from 30 days after the onset of symptoms of COVID-19 without risk of dissemination.

In persistent hyposmia other than chronic rhinosinusitis, the only treatment that has proven its efficacy is nasal irrigation associated with budesonide and olfactory rehabilitation. However, this drug does not have marketing authorisation in France for this indication.

DETAILED DESCRIPTION:
This is a multicenter randomized trial to evaluate the efficacy of local budesonide (nasal irrigation) in the management of persistent hyposmia in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age;
* Patient with a suspected SARS-CoV-2 infection in a epidemic context, whether or not confirmed by PCR, or contact close to a PCR-confirmed case, typical chest CT scan (unsystematized frosted glass areas predominantly sub-pleural, and at a later stage of alveolar condensation with no excavations neither nodules nor masses) or positive serology ;
* Patient with isolated acute hyposmia persisting at D30. of the onset of signs of CA-MRSA-CoV-2 infection;
* Absence of PCR-confirmed SARS-CoV-2 portage at the time of inclusion

Exclusion Criteria:

* Known hypersensitivity to budesonide or to any of the excipients of the medicine;
* Hemostasis disorder, or epistaxis;
* Oromo-oral-nasal and ophthalmic herpes virus infection;
* Long-term corticosteroid treatment;
* Treatment with potent CYP3A4 inhibitors (e.g., CYP3A4 inhibitors); ketoconazole, itraconazole, voriconazole, posaconazole, clarithromycin, telithromycin, nefazodone and HIV proteases) ;
* Forms of CoV-2-SARS with respiratory signs or other than anosmia persisting at 30 days from the onset of symptoms;
* Hyposmia persisting for more than 90 days after onset of symptoms;
* Other causes of hyposmia revealed on interrogation or an MRI;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Patient with more than 2 points on the ODORATEST | 30 days
  Percentage of patients with an improvement of more than 2 points on the ODORATEST score (5) after 30 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mary DAVAL, Principal Investigator — Hopital Fondation A de Rothschild
Locations (1):
- Amélie YAvchitz, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hautefort C, Corre A, Poillon G, Jourdaine C, Housset J, Eliezer M, Verillaud B, Slama D, Ayache D, Herman P, Yavchitz A, Guillaume J, Herve C, Bakkouri WE, Salmon D, Daval M. Local budesonide therapy in the management of persistent hyposmia in suspected non-severe COVID-19 patients: Results of a randomized controlled trial. Int J Infect Dis. 2023 Nov;136:70-76. doi: 10.1016/j.ijid.2023.08.022. Epub 2023 Aug 29. PMID 37652094
- [Derived] Daval M, Corre A, Palpacuer C, Housset J, Poillon G, Eliezer M, Verillaud B, Slama D, Ayache D, Herman P, Jourdaine C, Herve C, El Bakkouri W, Salmon D, Hautefort C. Efficacy of local budesonide therapy in the management of persistent hyposmia in COVID-19 patients without signs of severity: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Jul 20;21(1):666. doi: 10.1186/s13063-020-04585-8. PMID 32690074